CLINICAL TRIAL: NCT07089381
Title: Efficacy and Safety of Resveratrol in Patients With Rheumatoid Arthritis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rana El-Dash, Assistant Lecturer/Pharmacist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 338
Record Dates: First submitted 2025-07-21; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Rheumatic Arthritis; Rheumatoid Arthritis (RA) Prevention; Inflamation; Antioxidant; Anti Oxidative Stress; Anti Aging; C Reactive Protein; Methotrexate; Quality of Life Outcomes
MeSH Terms: conditions — Rheumatic Fever; Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol group (Experimental): 59 patients will receive the standard treatment for management of RA in addition to Resveratrol 1 gm daily for three month daily.
  Interventions: Dietary Supplement: Resveratrol 1 gm.
- Control arm (Active Comparator): 59 patients will receive the standard treatment for management of RA for 3 months.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Dietary Supplement: Resveratrol 1 gm. — 59 patients will receive the standard treatment for management of RA in addition to Resveratrol 1 gm daily, (Organix, Egypt) (given as one 1000 mg tablets once daily) for 3 months.
  Arms: Resveratrol group
Drug: Methotrexate — 59 patients will receive the standard treatment for management of RA for 3 months
  Arms: Control arm

SUMMARY:
The aim of the current study is to evaluate the effects of resveratrol on the clinical outcome(s) of patients with moderate rheumatoid arthritis.

Objectives :

1. To investigate the effects of Resveratrol on inflammation and oxidative stress by measuring:

   * Serum Sirtuin 1(SIRT1)
   * Serum Myeloperoxidase (MPO)
   * Serum C-reactive protein (CRP)
2. To investigate the effects of Resveratrol on disease activity by measuring the disease activity (DAS28 score).
3. To investigate the effect of Resveratrol on improving the quality of life using the Health Assessment Questionnaire Disability index (HAQ-DI).
4. To assess any adverse effects related to Resveratrol.

Patients:

Eligible patients (no=118) will be randomly assigned in a 1:1 ratio to one of two groups:

1. Control group: 59 patients will receive the standard treatment for management of RA for 3 months.
2. Resveratrol group: 59 patients will receive the standard treatment for management of RA in addition to Resveratrol 1 gm daily, (Organix Egypt) (given as one 1000 mg tablets once daily) for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years old
* Established diagnosis of RA according to American College of Rheumatology/European league Against Rheumatism (ACR/EULAR) 2010 criteria (Aletaha et al., 2010), presented with moderate to high disease activity identified as disease activity score-28 based on C-reactive protein (CRP) levels (DAS-28-CRP) >3.2.
* Patients receiving stable regimen of one or more csDMARDs for at least the past 3 months.
* RA Patients with Moderate or high disease activity identified as disease activity score-28 based on C-reactive protein (CRP) levels (DAS-28-CRP) >3.2.

Exclusion Criteria:

* Patients receiving biologic DMARDs therapy for RA
* Patients taking any other anti-inflammatory drugs
* Patients taking any other antioxidants
* Pregnant and lactating women
* Other rheumatological, inflammatory diseases or malignancies
* Smokers
* Thyroid illnesses
* Patients with impaired liver functions (liver transaminases level ≥ three times upper normal limits), impaired kidney functions (estimated glomerular filtration rate (eGFR) < 30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
To investigate the effects of Resveratrol on inflammation and oxidative stress by measuring: • Serum Sirtuin 1(SIRT1) • Serum Myeloperoxidase (MPO) • Serum C-reactive protein (CRP) | From 3 to 6 Months

SECONDARY OUTCOMES:
2. To investigate the effects of Resveratrol on disease activity by measuring the disease activity (DAS28 score). | From 3 to 6 Months.
To investigate the effect of Resveratrol on improving the quality of life using the Health Assessment Questionnaire Disability index (HAQ-DI). | From 3 to 6 Months.

OTHER OUTCOMES:
To assess any adverse effects related to Resveratrol. | From 3 to 6 Months.

CONTACTS AND LOCATIONS:
Overall Officials: Lamia El-Wakeel, Professor of Clinical Pharmacy, Study Director — Clinical Pharmacy Department, Faculty of Pharmacy, Ain Shams University; Sarah Zaki, Professor of Clinical Pharmacy, Study Director — Clinical Pharmacy Departement, Faculty of Pharmacy, Ain Shams University; Al Shymaa Farouk, Lecturer of Internal Medicine, Study Chair — Rheumatology and Clinical Immunology, Faculty of Medicine, Ain Shams University; Rana El-Dash, Assistant Lecturer, Principal Investigator — Clinical Pharmacy Department, Faculty of Pharmacy, Ain Shams University
Locations (1):
- Department of Rheumatology at Ain Shams university hospital, Cairo, Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang G, Xie X, Yuan L, Qiu J, Duan W, Xu B, Chen X. Resveratrol ameliorates rheumatoid arthritis via activation of SIRT1-Nrf2 signaling pathway. Biofactors. 2020 May;46(3):441-453. doi: 10.1002/biof.1599. Epub 2019 Dec 28. PMID 31883358
- [Background] Kciuk M, Garg A, Rohilla M, Chaudhary R, Dhankhar S, Dhiman S, Bansal S, Saini M, Singh TG, Chauhan S, Mujwar S, Gielecinska A, Kontek R. Therapeutic Potential of Plant-Derived Compounds and Plant Extracts in Rheumatoid Arthritis-Comprehensive Review. Antioxidants (Basel). 2024 Jun 27;13(7):775. doi: 10.3390/antiox13070775. PMID 39061843
- [Background] Mousavi SE, Nejadghaderi SA, Khabbazi A, Alizadeh M, Sullman MJM, Kaufman JS, Collins GS, Safiri S. The burden of rheumatoid arthritis in the Middle East and North Africa region, 1990-2019. Sci Rep. 2022 Nov 11;12(1):19297. doi: 10.1038/s41598-022-22310-0. PMID 36369238
- [Background] Poniewierska-Baran A, Bochniak O, Warias P, Pawlik A. Role of Sirtuins in the Pathogenesis of Rheumatoid Arthritis. Int J Mol Sci. 2023 Jan 12;24(2):1532. doi: 10.3390/ijms24021532. PMID 36675041
- [Background] Diab A, Omar A, Maaty A, Abdalla M. Plasma and Synovial Fluid Levels of Myeloperoxidase in Patients with Rheumatoid Arthritis and Its Correlation with Disease Activity. Suez Canal University Medical Journal. 2023;26(2):0-0. doi:10.21608/scumj.2023.304689
- [Background] Garcia-Martinez BI, Ruiz-Ramos M, Pedraza-Chaverri J, Santiago-Osorio E, Mendoza-Nunez VM. Effect of Resveratrol on Markers of Oxidative Stress and Sirtuin 1 in Elderly Adults with Type 2 Diabetes. Int J Mol Sci. 2023 Apr 18;24(8):7422. doi: 10.3390/ijms24087422. PMID 37108584
- [Background] Oliveira ALB, Monteiro VVS, Navegantes-Lima KC, Reis JF, Gomes RS, Rodrigues DVS, Gaspar SLF, Monteiro MC. Resveratrol Role in Autoimmune Disease-A Mini-Review. Nutrients. 2017 Dec 1;9(12):1306. doi: 10.3390/nu9121306. PMID 29194364
- [Background] Khojah HM, Ahmed S, Abdel-Rahman MS, Elhakeim EH. Resveratrol as an effective adjuvant therapy in the management of rheumatoid arthritis: a clinical study. Clin Rheumatol. 2018 Aug;37(8):2035-2042. doi: 10.1007/s10067-018-4080-8. Epub 2018 Apr 3. PMID 29611086